CLINICAL TRIAL: NCT03859635
Title: Randomized Prospective Study Comparing Exparel Erector Spinae Plane Block vs Simple Bupivacaine Erector Spinae Plane Block vs Exparel Surgeon Infiltration for Postoperative Analgesia Following Video-assisted Thoracoscopic Surgery
Brief Title: Erector Spinae Block Versus Surgeon Infiltration in VATS Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Yar Yeap, Assistant Professor of Clinical Anesthesiology. Director, Acute Pain Service, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1809656804
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative; Thoracic; Acute Pain
Keywords: acute pain; VATS
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Patients are randomized into one of three groups:
  1. Ultrasound guided LB Erector Spinae Plane Block with 20ml of Exparel and 10ml 0.25% bupivacaine
  2. Ultrasound guided SB Erector Spinae Plane Block with 30ml 0.5% bupivacaine
  3. Surgeon Infiltration under video guidance with 20ml of Exparel and 10ml of 0.25% bupivacaine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ultrasound guided Liposomal Bupivacaine Erector Spinae Block (Active Comparator): All the erector spinae plane blocks will be placed preoperatively using Liposomal Buvicaine. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service or the attending anesthesiologist in the operating room.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine, 0.25%
- Ultrasound guided Standard Bupivacaine Erector Spinae Block (Active Comparator): All the erector spinae plane blocks will be placed preoperatively using Liposomal Buvicaine. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service or the attending anesthesiologist in the operating room.
  Interventions: Drug: Bupivacaine, 0.5%
- Surgeon Infiltration (Active Comparator): At the end of the surgery, the surgeon will infiltrate liposomal bupivacaine under thoracoscopic guidance along the intercostal nerves from T4-T8.
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine, 0.25%

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 20 ml
  Arms: Surgeon Infiltration; Ultrasound guided Liposomal Bupivacaine Erector Spinae Block
Drug: Bupivacaine, 0.25% — 10 ml
  Arms: Surgeon Infiltration; Ultrasound guided Liposomal Bupivacaine Erector Spinae Block
Drug: Bupivacaine, 0.5% — 30 ml
  Arms: Ultrasound guided Standard Bupivacaine Erector Spinae Block

SUMMARY:
The study is comparing the difference between erector spinae block and surgeon infiltration after VATS (Video Assisted Thoracoscopic Surgery). The outcomes measured are pain scores, opioid usage, opioid side effects, and patient satisfaction.We are also also studying the effectiveness of liposomal bupivacaine (EXPAREL) in a block by randomizing patients to both EXPAREL erector spinae block and simple bupivacaine erector spinae block.

DETAILED DESCRIPTION:
A total of 120 subjects will be randomized by a computer program into three groups (40 per group): The primary investigator will inform the anesthesiologist who will be doing the block as to what group the patients are randomized to. The research staff completing the patients assessments will be blinded to the randomization.

For the LB group (Ultrasound guided LB Erector Spinae Plane Block), patients should receive a total of 10ml 0.25% bupivacaine plus 20ml Exparel® (15ml at T4 and 15ml at T8) For the SB group (Ultrasound guided SB Erector Spinae Plane Block), patients should receive a total of 30ml 0.5% bupivacaine. (15ml at T4 and 15ml at T8) For the SI group (under video guidance) injected by surgeon using 10ml 0.25% bupivacaine plus 20ml Exparel

All the erector spinae plane blocks will be placed preoperatively after sedation, before intubation and prior to surgery. All procedures will be placed under the supervision of the attending anesthesiologist on the acute pain service or the attending anesthesiologist in the operating room.

For the ESP block, an ultrasound probe is used to visualize the ES musculature about 3 cm laterally from the spinous process. In a cephalad-to-caudad direction advance the needle and inject the anesthetic in the interfacial plane deep to the ES muscles. Confirm positioning by visualization of needle tip and elevation of ES muscles off the transverse process with anesthetic injection. Injection will be performed at T4 and T8 level.

Surgeon infiltration is performed intraoperatively under direct thoracoscopic guidance. The intercostal space will be visualized and injected with LB. Typically, T4 through T8 are infiltrated with the anesthetic mixture.

All patients will be placed on ERAS protocol, which is our standard of practice.

Opioid usage after the block will be recorded by a member of the research team. Pain scores at rest and on movement (knee flexion) will be measured by the investigator using Visual Analog Scale (VAS). Nausea will be measured using a categorical scoring system (none=0; mild=1; moderate=2; severe=3). Sedation scores will also be assessed by a member of the study team using a sedation scale (awake and alert=0; quietly awake=1; asleep but easily roused=2; deep sleep=3). All these parameters will be measured at 1, 24, 48 and 72 hours after the surgery.

All patients will receive a phone call 6 months after surgery for assessment for chronic post-surgical pain. Patients will be assessed by a member of the research team over the phone. They will be assessed on their pain score and narcotic usage by using the Brief Pain Inventory. Study participation will conclude after the 6 month follow questionnaire has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Pt undergoing VATS including but not limited to wedge or lobectomy at Indiana University Hospital
* ASA 1,2,3 or 4
* Age 18 or older, male or female
* Desires regional anesthesia for postoperative pain control

Exclusion criteria:

* Any contraindication for Erector Spinae Plane block
* History of substance abuse in the past 6 months which would include heroin, marijuana or any other illegal street drugs
* Patient staying intubated after surgery
* Patient (home dose) taking more than 30mg PO morphine equivalent per day
* Known allergy or other contraindications to the study medications, which include dilaudid and bupivacaine.
* Pts. scheduled for a pleurodesis, decortication or esophagectomy at Indiana University Hospital

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2022-11-06 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yar Yeap, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bottiger BA, Esper SA, Stafford-Smith M. Pain management strategies for thoracotomy and thoracic pain syndromes. Semin Cardiothorac Vasc Anesth. 2014 Mar;18(1):45-56. doi: 10.1177/1089253213514484. Epub 2013 Dec 12. PMID 24336691
- [Background] Singh S, Chowdhary NK. Erector spinae plane block an effective block for post-operative analgesia in modified radical mastectomy. Indian J Anaesth. 2018 Feb;62(2):148-150. doi: 10.4103/ija.IJA_726_17. No abstract available. PMID 29491525
- [Background] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392
- [Background] Rao Kadam V, Currie J. Ultrasound-guided continuous erector spinae plane block for postoperative analgesia in video-assisted thoracotomy. Anaesth Intensive Care. 2018 Mar;46(2):243-245. No abstract available. PMID 29519230
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Taylor R, Massey S, Stuart-Smith K. Postoperative analgesia in video-assisted thoracoscopy: the role of intercostal blockade. J Cardiothorac Vasc Anesth. 2004 Jun;18(3):317-21. doi: 10.1053/j.jvca.2004.03.012. PMID 15232812
- [Background] Wu ZQ, Min JK, Wang D, Yuan YJ, Li H. Liposome bupivacaine for pain control after total knee arthroplasty: a meta-analysis. J Orthop Surg Res. 2016 Jul 22;11(1):84. doi: 10.1186/s13018-016-0420-z. PMID 27443874
- [Background] Yu ZX, Yang ZZ, Yao LL. Effectiveness of liposome bupivacaine for postoperative pain control in total knee arthroplasty: A PRISMA-compliant meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Mar;97(13):e0171. doi: 10.1097/MD.0000000000010171. PMID 29595645
- [Background] Ma TT, Wang YH, Jiang YF, Peng CB, Yan C, Liu ZG, Xu WX. Liposomal bupivacaine versus traditional bupivacaine for pain control after total hip arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jun;96(25):e7190. doi: 10.1097/MD.0000000000007190. PMID 28640101
- [Background] Raman S, Lin M, Krishnan N. Systematic review and meta-analysis of the efficacy of liposomal bupivacaine in colorectal resections. J Drug Assess. 2018 Jun 29;7(1):43-50. doi: 10.1080/21556660.2018.1487445. eCollection 2018. PMID 29988796
- [Background] Knudson RA, Dunlavy PW, Franko J, Raman SR, Kraemer SR. Effectiveness of Liposomal Bupivacaine in Colorectal Surgery: A Pragmatic Nonsponsored Prospective Randomized Double Blinded Trial in a Community Hospital. Dis Colon Rectum. 2016 Sep;59(9):862-9. doi: 10.1097/DCR.0000000000000648. PMID 27505115
- [Background] Knight RB, Walker PW, Keegan KA, Overholser SM, Baumgartner TS, Ebertowski JS 2nd, Aden JK, White MA. A Randomized Controlled Trial for Pain Control in Laparoscopic Urologic Surgery: 0.25% Bupivacaine Versus Long-Acting Liposomal Bupivacaine. J Endourol. 2015 Sep;29(9):1019-24. doi: 10.1089/end.2014.0769. Epub 2015 Jun 5. PMID 25897552
- [Background] Noviasky J, Pierce DP, Whalen K, Guharoy R, Hildreth K. Bupivacaine liposomal versus bupivacaine: comparative review. Hosp Pharm. 2014 Jun;49(6):539-43. doi: 10.1310/hpj4906-539. PMID 24958971
- [Result] Kaplowitz J, Papadakos PJ. Acute pain management for video-assisted thoracoscopic surgery: an update. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):312-21. doi: 10.1053/j.jvca.2011.04.010. Epub 2011 Jun 25. No abstract available. PMID 21705236

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Started | 40 | 40 | 40
Completed | 37 | 35 | 33
Not Completed | 3 | 5 | 7

BASELINE CHARACTERISTICS:
Population: Total of 120 patients consented for the study. 15 patients were excluded from the study, leaving a total of 105 patients at study completion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration | Total
Number analyzed (Participants) | 37 | 35 | 33 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9) | 64 (10) | 66 (12) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 26 | 15 | 60
  Male | 18 | 9 | 18 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: weight in kg] | 76.44 (19.02) | 79.59 (16.11) | 86.19 (15.33) | 80.56 (17.29)
BMI [Mean (Standard Deviation); unit: Body Mass Index in kg/m^2] | 25.90 (5.57) | 28.81 (4.72) | 29.89 (4.89) | 28.13 (5.32)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Study Will be 24 Hours VAS Pain Score at Rest
Description: The VAS score will be taken at rest using Visual Analog Scale (VAS). Using a scale of 0-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: 24 hours pain score at rest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
score on a scale | 4.1 (2.5) | 4.3 (2.6) | 3.3 (2.3)

2. Primary Outcome: The Primary Endpoint of This Study Will be 24 Hours VAS Pain Score With Movement
Description: The VAS score will be taken after movement (knee flexion) using Visual Analog Scale (VAS). Using a scale of 0-10 for documentation with 10 being the worst pain and 0 being no pain
Time Frame: 24 hours pain score with movement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
score on a scale | 6.0 (2.8) | 6.3 (2.3) | 4.5 (2.9)

3. Primary Outcome: The Primary Endpoint of This Study Will be 48 Hours VAS Pain Score at Rest
Description: as for outcome 1
Time Frame: 48 hours pain score at rest
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
score on a scale | 3.1 (2.3) | 3.4 (2.5) | 2.8 (2.1)

4. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 72 Hours
Description: Opioid consumption between 48-72hr will be collected by a study team member per protocol time requirements
Time Frame: Opioid consumption will be measured at 72 hours post op. The total amount will be recorded.]
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalant/day
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
mg morphine equivalant/day | 26 [18 to 68] | 48 [28 to 72] | 40 [20 to 136]

5. Secondary Outcome: Average Nausea Scores Over 72 Hours
Description: Nausea scores will be collected by a study team member post operatively up to 3 days per protocol. Nausea will be recorded as None=0, Mild=1, Moderate=2, Severe=3.
Time Frame: Nausea scores will be documented at 1 hour post op, 24,48,and 72 hours after the block. The scores will then be averaged
Population: as for baseline characteristics
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
units on a scale | 0.14 [0 to 3] | 0.14 [0 to 2] | 0.06 [0 to 2]

6. Secondary Outcome: Average Sedation Scores Over 72 Hours
Description: Sedation scores will be documented by a study team member post operatively up to 3 days per protocol requirements. Determining if patient is Awake/Alert=0, Quietly Awake=1, Asleep but Arousable=2, or Deep Sleep=3
Time Frame: Sedation scores will be documented at 1 hour post op, 24,48,and 72 hours after the block. The scores will then be averaged.]
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
units on a scale | 0.08 [0 to 2] | 0.03 [0 to 1] | 0 [0 to 0]

7. Secondary Outcome: Subjects Overall Satisfaction Scores at Hour 24
Description: Subjects will be followed up at 24 hours post operatively by a study team member to document patient overall satisfaction scores. The scores are collected as Very Unsatisfied=0, Unsatisfied=1, Neutral=2, Satisfied=3, Very Satisfied=4
Time Frame: post operatively at hour 24
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
units on a scale | 3.5 [3 to 4] | 4 [1 to 4] | 3 [2 to 4]

8. Secondary Outcome: Subjects Overall Satisfaction Scores at Hour 48
Description: Subjects will be followed up at 48 hours post operatively by a study team member to document patient overall satisfaction scores. The scores are collected as Very Unsatisfied=0, Unsatisfied=1, Neutral=2, Satisfied=3, Very Satisfied=4
Time Frame: post operatively at hour 48
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
units on a scale | 3 [2 to 4] | 4 [1 to 4] | 4 [1 to 4]

9. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 48 Hours
Description: Opioid consumption at 24-48hr post op will be collected by a study team member per protocol time requirements
Time Frame: Opioid consumption will be measured at 48 hours post op. The total amount will be recorded.]
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalant/day
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
mg morphine equivalant/day | 48 [16 to 88] | 34 [22 to 76] | 60 [28 to 80]

10. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 24 Hours
Description: Opioid consumption at 1-24 hr postop will be collected by a study team member per protocol time requirements
Time Frame: Opioid consumption will be measured at 24 hours post op. The total amount will be recorded.]
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalant/day
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
mg morphine equivalant/day | 38 [18 to 62] | 40 [24 to 96] | 36 [20 to 68]

11. Secondary Outcome: Secondary Endpoint Includes Total Opioid Consumption at 1 Hour
Description: Opioid consumption at 1hr will be collected by a study team member per protocol time requirements
Time Frame: Opioid consumption will be measured at 1 hour post op. The total amount will be recorded.]
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: mg morphine equivalant
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
mg morphine equivalant | 16 [8 to 20] | 12 [8 to 20] | 8 [4 to 16]

12. Primary Outcome: The Primary Endpoint of This Study Will be 48 Hours VAS Pain Score With Movement
Description: as for outcome 2
Time Frame: 48 hours pain score with movement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ultrasound Guided Liposomal Bupivacaine Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
Number analyzed (Participants) | 37 | 35 | 33
score on a scale | 4.6 (2.6) | 5.3 (2.4) | 3.8 (2.6)

ADVERSE EVENTS:
Time Frame: Any adverse events from day of surgery til 6 months after surgery are documented..
Groups:
- Ultrasound Guided Loposomal Erector Spinae Block: Group 1-Ultrasound guided Liposomal Erector Spinae Block
- Ultrasound Guided Standard Bupivacaine Erector Spinae Block: Group-2-Ultrasound guided Standard Bupivacaine Erector Spinae Block
- Surgeon Infiltration: Group 3-Surgeon Infiltration
Arm/Group | Ultrasound Guided Loposomal Erector Spinae Block | Ultrasound Guided Standard Bupivacaine Erector Spinae Block | Surgeon Infiltration
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 1/37 | 0/35 | 1/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound Guided Loposomal Erector Spinae Block (N=37) | Ultrasound Guided Standard Bupivacaine Erector Spinae Block (N=35) | Surgeon Infiltration (N=33)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (33)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03859635/Prot_SAP_002.pdf